CLINICAL TRIAL: NCT05144490
Title: The Effect of Brief Bodyweight Exercise on Acute Glycemic Control in Healthy Inactive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: York University (Other)
Responsible Party: Principal Investigator, Martin Gibala, Professor, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 13864
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Exercise
Keywords: Glycemic Control
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bodyweight Exercise (Experimental): A standardized 11-minute bodyweight exercise session that involves a 1-minute warm-up followed by 5, 1-minute bouts of exercise at a self-selected "challenging" pace, interspersed with 1-minute periods of low-intensity exercise for recovery.
  Interventions: Other: Exercise
- Non-Exercise Control (No Intervention): An 11-minute period of quiet sitting.

INTERVENTIONS:
Other: Exercise — A single session of bodyweight exercise
  Arms: Bodyweight Exercise

SUMMARY:
This study will investigate whether an 11-minute bodyweight exercise session can improve short-term glycemic control. Glycemic control refers to the process of how the body regulates blood sugar. The process can be measured in different ways. This study will use a small device called a continuous glucose monitor to measure changes in glucose levels over a 24-hour period. Participants will complete two trials and the investigators will compare glycemic control after the exercise session and a control period that does not involve exercise. Food intake will be controlled such that each participant will consume the same diet in both conditions. This study will help determine whether a single session of bodyweight exercise affects glycemic control.

DETAILED DESCRIPTION:
This study will investigate whether an 11-minute bodyweight exercise session can improve short-term glycemic control. Glycemic control will be assessed using continuous glucose monitoring for 24 hours following exercise or a control condition that does not involve exercise. The exercise and control periods will be directly supervised by a study investigator. Participants will complete two trials in a randomized, crossover manner separated by 7 days. Food intake will be controlled such that each participant will consume the same diet over the 24-hour period of measurement in both conditions. Standardized meals will be provided to participants prior and following the exercise and control conditions. This study will determine whether a single session of bodyweight exercise affects glycemic control as primarily assessed by mean 24-hour glucose.

ELIGIBILITY:
Inclusion Criteria:

* Inactive, defined as not meeting the physical activity targets in the Canadian 24-Hour Movement Guidelines for Adults.
* Deemed able to safely participate in physical activity and exercise, as determined by the Canadian Society for Exercise Physiology (CSEP) Get Active Questionnaire prescreening tool.

Exclusion Criteria:

- Experiencing a condition that might preclude safe participation in physical activity and exercise, as determined by answering "Yes" to any question on Page 1 of the CSEP Get Active Questionnaire.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
24-hour mean glucose | 24-hour measurement period
  Mean glucose following the bodyweight exercise or control condition

SECONDARY OUTCOMES:
Glycemic variability | 24-hour measurement period
  Variability in glucose measured following exercise or control
Peak glucose | 2-hour measurement period after each meal
  Peak glucose measured after each meal following exercise or control
2-hour postprandial mean glucose | 2-hour measurement period after each meal
  Mean glucose measured after each meal following exercise or control

CONTACTS AND LOCATIONS:
Overall Officials: Martin Gibala, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No